CLINICAL TRIAL: NCT06641557
Title: A Phase I, 7-Day Dosing Study of 200 Mg IkT-148009 to Determine the Safety, Tolerability and Pharmacokinetics (PK) of IkT-148009 in Older Adult and Elderly Healthy Volunteers
Brief Title: A Phase I Dosing Study of IkT-148009.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ABLi Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IkT-148009-102
Record Dates: First submitted 2024-09-12; First posted 2024-10-15 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 200mg (Experimental): IkT-148009 will be administered as 4x50mg gelatin capsules
  Interventions: Drug: 200mg of Ikt-148009

INTERVENTIONS:
Drug: 200mg of Ikt-148009 — 4 50mg capsules

SUMMARY:
This is a Phase 1 study in older adult or elderly healthy volunteer subjects to measure the safety, tolerability and pharmacokinetic (PK) profile of IkT-148009 capsules given as multiple capsules.

DETAILED DESCRIPTION:
This is a Phase 1 study in older adult or elderly healthy volunteer subjects to measure the safety, tolerability and pharmacokinetic (PK) profile of IkT-148009 capsules given as multiple capsules.

This is a single arm study with subjects to treatment with IkT-148009 only. The study will consist of a total of up to 15 visits over a period of up to 29 days prior to dosing, 7 days of dosing and 14 days of follow up.

Subjects will receive a single daily dose of study drug with a meal for a period of up to 7 days. A full breakfast must be consumed prior to receiving the dose study drug. Subjects will be confined to the unit for approximately 12 days.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject must have all questions about the study answered and must have signed the informed consent document before any study-specific procedures are performed.

  2. Men or women aged 45 to 70 years at screening (both inclusive) of any race. 3. Subjects must be otherwise healthy and ambulatory, with no history or evidence of clinically relevant medical disorders 4. Mini Mental State Examination (MMSE) ≥ 28 5. Physical examination, clinical laboratory values, vital signs, and the electrocardiogram (ECGs) are clinically acceptable to the Investigator. Body weight ≥ 45 kg. Body Mass Index (BMI) ≥ 18 and ≤33 kg/m2.

  6. Female subjects must be postmenopausal or surgically sterile or sterile for other medical reason.

  7. Male subjects must agree to practice an acceptable method of highly effective birth control.

  8. Males must be willing to abstain from sperm donation from the screening visit, while on study and through 30 days after receiving the last dose of study drug.

Exclusion Criteria:

* 1. Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at the screening and admission visits.

  2. Clinically significant abnormal findings on physical examination or 12-lead electrocardiogram (ECG) at the screening or admission visits.

  3. Significant history (within six months prior to receiving the study drug) and/or presence of clinically significant medical, surgical or psychiatric disorder in the judgement of the investigator.

  4. History of clinically significant problems in the retina as reported by a subject

  5. eGFR < 60 mg/mL

  6. Creatinine, Amylase and/or Lipase > ULN

  7. Any malignancy in the 5 years prior to screening excluding basal cell carcinoma or squamous cell carcinoma of the skin or cervical carcinoma in situ that have been successfully treated.

  8. Any subject with a history, presence and/or current evidence of serologic positive result for hepatitis B surface antigen, hepatitis C antibodies, or HIV antibodies 1 or 2. Subjects considered to be cured for hepatitis C will be eligible.

  9. Recent history (within previous six months prior to screening) of alcohol or drug abuse (as judged by the investigator) or has consumed > 2 alcohol drinks/day during the last three months prior to screening.

  10. Any subject with known hypersensitivity to IkT-148009. 11. Donation of blood, plasma, or acute loss of blood within 60 days prior to screening visit.

  12. Use of tobacco or nicotine-containing products during the 60 days prior to screening and for the duration of the study.

  13. Any subject who has received treatment with an investigational drug during the 30 days prior to screening.

  14. Investigative site personnel or their immediate families (spouse, parent, child or sibling whether biological or legally adopted).

  15. Any subject unwilling or unable to comply with study procedures.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Participant Safety | Through study completion, an average of 50 days
  Adverse event reporting
Participant Safety - vital signs | Through study completion, an average of 50 days
  Changes in vital sign measurements including HR and blood pressure.
Participant Safety - clinical lab values | Through study completion, an average of 50 days
  Changes in clinical laboratory data consisting of CBC, Serum Chemistry, FSH.
Participant Safety | Through study completion, an average of 50 days
  Electrocardiogram [ECG] parameters of ventricular rate, RR or PR interval, QRS complex, and QTcF interval.
Participant Safety | Through study completion, an average of 50 days
  C-SSRS assessment values.
Participant Tolerability | Through study completion, an average of 50 days
  Percent completers
Assess the pharmacokinetics (PK) of IkT-148009 | Through study completion, an average of 50 days
  Pharmacokinetic parameters:
  • Area under the concentration-time curve from time zero to 96 hours (AUC0-∞)
Assess the pharmacokinetics (PK) of IkT-148009 | Through study completion, an average of 50 days
  Pharmacokinetic parameters:
  • Maximum plasma concentration (Cmax)
Assess the pharmacokinetics (PK) of IkT-148009 | Through study completion, an average of 50 days
  Pharmacokinetic parameters:
  • Area under the concentration-time curve from time zero to last time point (AUC0-last)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No